CLINICAL TRIAL: NCT02345616
Title: Role of the Nitric Oxide (NO) in Pre-oxygenation Before Anesthetic Induction in Patients With a Pulmonary Hypertension in Cardiac Surgery. Pilot Study of Feasibility
Acronym: NOCaPH
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: ARAMU Association (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHU-0221; 2014-003338-15 (EudraCT Number)
Record Dates: First submitted 2015-01-20; First posted 2015-01-26 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Pulmonary Hypertension
Keywords: Cardiac surgery; Pulmonary hypertension; Nitric oxide; Induction anesthesia
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Nitric Oxide

ARMS (1):
- Nitric oxyde (Experimental)
  Interventions: Drug: Nitric oxide

INTERVENTIONS:
Drug: Nitric oxide

SUMMARY:
The pulmonary hypertension (HTP) due to a left heart disease or a hypoxemiant lung disease is frequent in cardiac surgery. The HTP represents an independent risk factor of morbidity and mortality in cardiac surgery, entering to the criteria of Euroscore evaluation (European System for Cardiac Operative Risk Evaluation).

An acute perioperative hemodynamic decompensation of these patients is frequent. Perioperative hemodynamic modifications, hypoxemia, hypercapnia, sympathetic stimulation, increase pulmonary vascular resistances (RVP) and might provoke right ventricular failure.

The anesthetic induction and the beginning of mechanical ventilation are the most sensible times due to the risk of hemodynamic decompensation. The suppression of the sympathetic tonus which is consequence of the anesthetic induction, decrease the systemic vascular resistances and lead to decrease of blood pressure. In return, the anesthetic induction is associated with an increase of pulmonary vascular resistances, resulting in increase of the postcharge and the work of the right ventricle (VD). These systemic and pulmonary hemodynamic modifications can lead to equalization, or even an inversion of the systemic and pulmonary pressures. As consequence, a hemodynamic collapse or even a heart arrest can arise.

The patients suffering from HTP are hypoxemic. They have very limited oxygen reserves due to decrease of the functional residual capacity (CRF). The apnea period, which follows the anesthetic induction, is often associated with a fast desaturation, even if a good pre-oxygenation was performed before. This desaturation causes an increase of the pulmonary vascular resistances with the hemodynamic consequences previously mentioned. A risk of hypoxic heart arrest is also present.

Nitric Oxide (NO) is an endogenous mediator produced from the vascular endothelium. The NO is a powerful vasodilator and is used in intensive care in inhaled way as selective pulmonary vasodilator (iNO). NO decreases the RVP, the shunt effect and improves the oxygenation by optimization of ventilation-perfusion ratio. The short lifetime of iNO (6sec approximately) allows a fast metabolism without inducing any undesirable effects such as the systemic hypotension.

No studies, until now, have investigated the use of iNO in pre-oxygenation before anesthetic induction in cardiac surgery.

We hope to demonstrate that iNO used in oxygenation before anesthetic induction will have a beneficial effect on the respiratory and cardiovascular parameters.

Our objective is to estimate the feasibility and the tolerance of iNO before anesthetic induction of the patients with a moderate or severe HTP programmed for cardiac surgery with extracorporeal circulation. The effect will be estimated in terms of efficiency (hemodynamic and respiratory optimization).

DETAILED DESCRIPTION:
Before the anesthetic induction every included patient will follow these protocol:

* Standard monitoring (ECG Electrocardiogram, SpO2 Pulsed oxygen saturation)
* Insertion of radial arterial line and periferic IV line under local anesthesia,
* Insertion of a internal jugular central line and Swan Ganz catheter under local anesthesia
* Preoxygenation in 100% oxygen for 10 min
* Further preoxygenation with a mixture of 100% oxygen associated with the iNO in a dose of 1,2 L / mn.
* Anesthesia induction and initiation of mechanical ventilation.
* Progressive decrease of iNO dose and stop of iNO administration.

ELIGIBILITY:
Inclusion Criteria:

- Age > 18 years old

* Open-heart cardiac surgery
* HTP Pulmonary hypertension (class 2 or 3) with PAPs (Systolic pulmonary artery pressure) > 40 mmHg diagnosed by preoperative righ cardiac catheterization or by transthoracic echocardiography.
* Patient have signed their consent according to the modalities described by the Code of Public health system.
* Patients affiliated to a national insurance (social security) system.

Exclusion Criteria:

* Heart transplant
* HTP of type 1, 4, 5 according to the classification of Dana Point(2008)
* Deficit in methemoglobin reductase
* Protocole refuse from patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-02; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Pulmonary arterial systolic, diastolic and mean pressure | at day 1
  These measures will be taken each minute between t0 (conditioning of the patient's arrival in the operating room) and the time when FiO2 (Fraction of inspired oxygen) will be 60% (when the endotracheal tube is in place, between 30 and 40 minutes after t0)
Pulmonary arterial mean/arterial mean ratio | at day 1
  These measures will be taken each minute between t0 (conditioning of the patient's arrival in the operating room) and the time when FiO2 (Fraction of inspired oxygen) will be 60% (when the endotracheal tube is in place, between 30 and 40 minutes after t0)
SpO2 (Pulsed oxygen saturation) | at day 1
  These measures will be taken each minute between t0 (conditioning of the patient's arrival in the operating room) and the time when FiO2 (Fraction of inspired oxygen) will be 60% (when the endotracheal tube is in place, between 30 and 40 minutes after t0)
FeO2 (Fraction expired oxygen) (data not available just during intubation phase) | at day 1
  These measures will be taken each minute between t0 (conditioning of the patient's arrival in the operating room) and the time when FiO2 (Fraction of inspired oxygen) will be 60% (when the endotracheal tube is in place, between 30 and 40 minutes after t0)
Cardiac index | at day 1
  These measures will be taken each minute between t0 (conditioning of the patient's arrival in the operating room) and the time when FiO2 (Fraction of inspired oxygen) will be 60% (when the endotracheal tube is in place, between 30 and 40 minutes after t0)
Systemic vascular resistances | at day 1
  These measures will be taken each minute between t0 (conditioning of the patient's arrival in the operating room) and the time when FiO2 (Fraction of inspired oxygen) will be 60% (when the endotracheal tube is in place, between 30 and 40 minutes after t0)
SVO2 (Central Venous Saturation) | at day 1
  These measures will be taken each minute between t0 (conditioning of the patient's arrival in the operating room) and the time when FiO2 (Fraction of inspired oxygen) will be 60% (when the endotracheal tube is in place, between 30 and 40 minutes after t0)
Sat O2 (Blood oxygen saturation) | at day 1
  These measures will be taken each minute between t0 (conditioning of the patient's arrival in the operating room) and the time when FiO2 (Fraction of inspired oxygen) will be 60% (when the endotracheal tube is in place, between 30 and 40 minutes after t0)
PaO2 (Partial pressure of arterial oxygen) | at day 1
  These measures will be taken each minute between t0 (conditioning of the patient's arrival in the operating room) and the time when FiO2 (Fraction of inspired oxygen) will be 60% (when the endotracheal tube is in place, between 30 and 40 minutes after t0)
MetHb (methemoglobin) | at day 1
  These measures will be taken each minute between t0 (conditioning of the patient's arrival in the operating room) and the time when FiO2 (Fraction of inspired oxygen) will be 60% (when the endotracheal tube is in place, between 30 and 40 minutes after t0)

SECONDARY OUTCOMES:
Systolic, diastolic and mean arterial pressure | at day 1
  These measures will be taken each minute between t0 (conditioning of the patient's arrival in the operating room) and the time when FiO2 will be 60% (when the endotracheal tube is in place, between 30 and 40 minutes after t0)

CONTACTS AND LOCATIONS:
Overall Officials: Vedat ELJEZI, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France